CLINICAL TRIAL: NCT03540849
Title: Maintenance Brentuximab Vedotin (Bv) Following Allogeneic Stem Cell Transplantation for Hodgkin Lymphoma Patient: A Prospective, Multicenter, Phase II Study.
Brief Title: BV After Allogeneic Hematopoietic Stem Cell Transplantation
Acronym: BV-ALLO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-122
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BV after allogeneic hematopoietic stem cell transplantation (Experimental)
  Interventions: Drug: Brentuximab Vedotin (Bv)

INTERVENTIONS:
Drug: Brentuximab Vedotin (Bv) — HL patients who are eligible for the study, will receive maintenance Bv. The first Bv dosage will be administered three months after allo-SCT (day 90) at the dosage of 1.8 mg/kg every 21 days for 12 cycles. post allo-SCT maintenance Bv for Hodgkin lymphoma

SUMMARY:
Despite a high recovery rate with chemotherapy and radiation therapy treatment, 15 to 30% of patients suffering from Hodgkin lymphoma are refractory or relapsed. Standard rescue treatment for these patients is chemotherapy followed by a hematopoietic stem cell auto-SCT. Despite a very good rate of complete sustainable response in 50% of the patients, another 50% of the patients relapse after increased therapy and require additional treatment. Consequently, one option for these patients is to offer a novel rescue therapy, enabling them to have partial or complete response, and offer them a hematopoietic stem cell allo-SCT. In the only prospective phase 2 study published by Sureda et al. assessing this therapeutic approach, the rate of mortality not linked to relapse was 8% at 100 days and 15% at 1 year. The progression-free survival rate was 48% at 1 year and 24% at 4 years. Relapse occurred between 3 and 35 months with a median of 6 months in 51% of the patients out of a total of 78 patients. Cumulative incidence of relapse was 37% at 1 year and 59% at 5 years.

Brentuximab Vedotin (Bv) is an anti-CD30 antibody-drug conjugate. This drug has shown its efficacy with very acceptable toxicity in patients suffering from advanced-stage Hodgkin lymphoma. Bv was consolidatively evaluated after an auto-SCT. 329 patients, at high risk of relapse after auto-SCT, received Bv (n=165) in a dose of 1.8 mg/kg every 3 weeks or a placebo (n=164) for 16 cycles. The progression-free survival median (validated by a panel of independent experts) was 42.9 months (95% CI 30,4-42 ; 9) for patients in the Bv group and 24.1 months (11.5 not reached) in the placebo group.

The purpose of our study is to reduce relapse rate by carrying out maintenance with Bv after allografting hematopoietic stem cells in a population of patients suffering from Hodgkin lymphoma with high risk of relapse after auto-SCT. Fifty eight patients have been slated for inclusion over a period of 2 years.

This is an open-label, prospective, multicenter, phase II trial consisting of post allo-SCT maintenance Bv for Hodgkin lymphoma.

Patients will be recruited over 24 months and be followed for 3 years after allo-SCT.

A total of 58 patients will be included in the study. The duration of the treatment period is approximately 10.7 months for 12 cycles of Bv.

End of study: end of study is defined by the last visit planned by the protocol of the last patient in follow-up, which means 3 years after allo-SCT.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged less than 18 or more than 65 years
2. Patients who received allo-SCT for relapse after autologous transplantation for Hodgkin's lymphoma
3. Patients who received tandem autologous and allogeneic stem cell transplantation for HL are eligible
4. Histologically confirmed CD30+ classical Hodgkin lymphoma according to local pathologist (excluding nodular lymphocyte predominant subtype)
5. Patients with Ann Arbor stage II-III or IV or extranodal localization at relapse post ASCT
6. Patients who previously received Bv may be included if the duration of response to initial Bv treatment is more than 3 months
7. Patients who previously received anti-PD1 drugs can be included
8. Voluntary written informed consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
9. Patients must be covered by a social security system
10. Female patients is either post-menopausal for at least 1 year before the screening visit or surgically sterile or if of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 6 months after the last dose of study drug
11. Male patients, even if surgically sterilized, (i.e., status post vasectomy) agree to practice effective barrier contraception during the entire study period and through 6 months after the last dose of study drug.
12. Performance status less or equal to 2

Exclusion Criteria:

1. Patients with histologically confirmed nodular lymphocyte predominant subtype
2. Female patient who are both lactating and breast-feeding or have a positive serum pregnancy test during the screening period or a positive pregnancy test on Day 1 before first dose of study drug
3. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to the protocol.
4. Known cerebral or meningeal disease (HL or any other etiology), including signs or symptoms of PML
5. Unstable diabetes mellitus (to avoid uninterpretable FDG-PET scan).
6. Symptomatic neurologic disease compromising normal activities of daily living or requiring medications
7. Any sensory or motor peripheral neuropathy greater than or equal to Grade 2
8. Known history of any of the following cardiovascular conditions

   Myocardial infarction within 2 years of enrollment :
   * New York Heart Association (NYHA) Class III or IV heart failure
   * Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure (CHF), angina, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
   * Recent evidence (within 6 months before first dose of study drug) of a left-ventricular ejection fraction less than 50%
9. Any active systemic viral, bacterial, or fungal infection requiring systemic antibiotics within 2 weeks prior to first study drug dose
10. Patients that have not completed any prior treatment chemotherapy and/or other investigational agents within at least 5 half-lives of last dose of that prior treatment
11. Known hypersensitivity to recombinant proteins, murine proteins, or to any excipient contained in the drug formulation of Bv.
12. Known human immunodeficiency virus (HIV) positive
13. Known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection
14. Diagnosed or treated for another malignancy within 3 years before the first dose or previously diagnosed with another malignancy and have evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
15. Patient who presented intolerance to Bv
16. Patient enrolled in other clinical research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2018-03-07 (Actual); Primary Completion 2020-03-07 (Estimated); Study Completion 2023-03-07 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of relapse (CIR) or progression at 12 months after allo-SCT | 12 month after allo-SCT

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No